CLINICAL TRIAL: NCT07395492
Title: Impact of App-Based Education and Low-Residue Diet Approaches on Colonoscopy Preparation in Naive Patients: A Randomized, Evaluator-Blind Controlled Trial
Brief Title: App-Based Education and Low-Residue Diet for Colonoscopy Preparation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Universal Integrated Corp. (Industry)
Responsible Party: Principal Investigator, Chen-Ming Hsu, Department of Gastroenterology and Hepatology, Chang Gung Memorial Hospital, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 202501149B0
Record Dates: First submitted 2025-12-17; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Bowel Preparation Solution
Keywords: Bowklean; Bowel preparation; Low-residue diet; boston bowel preparation scale

STUDY DESIGN:
Intervention Model Description: In this study, "naive patients" are defined as individuals who have never used Bowklean® as a bowel cleansing agent, or those who may have previously used other bowel preparation regimens but have not undergone any bowel cleansing procedure within the past three years. The Traditional Bowel Preparation approach consists of standard paper-based educational handouts and self-managed low-residue dietary restrictions. In contrast, the Advanced Bowel Preparation integrates a smartphone-based educational app (Tian Tian Yi Chi go, developed by UIC Corp.) with a Prepackaged Low-Residue Diet (PLD). The app provides timely reminders and interactive guidance, while PLD ensures dietary consistency and reduces errors arising from patient interpretation of dietary instructions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Bowel Preparation (No Intervention): The Traditional Bowel Preparation approach consists of standard paper-based educational handouts and self-managed low-residue dietary restrictions.
- Advanced Bowel Preparation (Experimental): Advanced Bowel Preparation integrates a smartphone-based educational app (Tian Tian Yi Chi go, developed by UIC Corp.) with a Prepackaged Low-Residue Diet (PLD).
  Interventions: Device: Tian Tian Yi Chi go APP (developed by UIC Corp); Dietary Supplement: Prepackaged Low-Residue Diet

INTERVENTIONS:
Device: Tian Tian Yi Chi go APP (developed by UIC Corp) — Bowl preparation educational app
  Arms: Advanced Bowel Preparation
Dietary Supplement: Prepackaged Low-Residue Diet — Prepackaged Low-Residue Diet
  Arms: Advanced Bowel Preparation

SUMMARY:
This prospective, randomized, evaluator-blind, parallel-group trial is designed to objectively compare the effectiveness of Advanced Bowel Preparation versus Traditional Bowel Preparation in patients undergoing colonoscopy. In this study, "naive patients" are defined as individuals who have never used Bowklean® as a bowel cleansing agent, or those who may have previously used other bowel preparation regimens but have not undergone any bowel cleansing procedure within the past three years. The Traditional Bowel Preparation approach consists of standard paper-based educational handouts and self-managed low residue dietary restrictions. In contrast, the Advanced Bowel Preparation integrates a smartphone based educational app with a Prepackaged Low-Residue Diet. All participants will use Bowklean®, a bowel preparation agent combining sodium picosulfate, magnesium oxide, and anhydrous citric acid.

The primary endpoint is the percentage of subjects that achieve adequate cleansing (score ≧ 6) in the Boston Bowel Preparation Scale (BBPS).

The secondary endpoints include the percentage of subjects that achieve excellent cleansing (score ≧ 8) in the BBPS, mean score in different colon segments (right, transverse, left), which are assessed with the BBPS, adenoma detection rate, sessile serrated polyp detection rate, and patient satisfaction.

DETAILED DESCRIPTION:
Bowel preparation is a important task for colonoscopy examination. Studies have demonstrated that using smartphone apps can improve patient compliance and the quality of bowel cleansing. Additionally, the use of prepackaged low residue diet (PLD) has become increasingly common. PLD are designed to minimize undigested food residue in the gut, facilitating a cleaner colon for procedures like colonoscopy. Implementing PLD can reduce the burden of dietary restrictions on patients and enhance the effectiveness of bowel preparation. This study aims to evaluate whether an advanced bowel preparation protocol that combines a smartphone application with a PLD can improve patient satisfaction, and the cleanliness of the colon compared to standard preparation methods.

This prospective, randomized, evaluator-blind, parallel-group trial is designed to objectively compare the effectiveness of Advanced Bowel Preparation versus Traditional Bowel Preparation in patients undergoing colonoscopy. In this study, "naive patients" are defined as individuals who have never used Bowklean® as a bowel cleansing agent, or those who may have previously used other bowel preparation regimens but have not undergone any bowel cleansing procedure within the past three years. The Traditional Bowel Preparation approach consists of standard paper-based educational handouts and self-managed low residue dietary restrictions. In contrast, the Advanced Bowel Preparation integrates a smartphone based educational app (Tian Tian Yi Chi go, developed by UIC Corp.) with a Prepackaged Low-Residue Diet (PLD). All participants will use Bowklean®, a bowel preparation agent combining sodium picosulfate, magnesium oxide, and anhydrous citric acid. Blinding of outcome evaluators (endoscopists) helps minimize assessment bias, while the randomized parallel-arm design supports robust group comparisons. This design allows a focused assessment of whether combining digital and dietary support can improve bowel cleanliness, detection outcomes, and patient satisfaction. Overall, this trial structure is intended to generate clinically relevant, real-world evidence on optimizing colonoscopy preparation by integrating pharmacologic, digital, and dietary strategies.

Primary Endpoint:

The percentage of subjects that achieve adequate cleansing (score ≧ 6) in the Boston Bowel Preparation Scale (BBPS).

The secondary endpoints include:

The percentage of subjects that achieve excellent cleansing (score ≧ 8) in the Boston Bowel Preparation Scale (BBPS).

Mean score in different colon segments (right, transverse, left), which are assessed with the BBPS.

Adenoma Detection Rate (ADR): Proportion of patients in whom at least one adenoma is detected during the colonoscopy.

Sessile Serrated Polyp (SSP) Detection Rate: Proportion of patients in whom at least one SSP is detected during the colonoscopy.

Patient Satisfaction: Satisfaction will be evaluated in three subcategories through a questionnaire:

1. Bowel cleansing agent: Assessing the experience and acceptability of using Bowklean.
2. Dietary restrictions: Evaluating satisfaction with the assigned low-residue dietary approach (PLD or self-prepared).
3. APP Satisfaction: For groups assigned to APP utilization, assessing the APP's ease of use, functionality, and perceived utility. 0800 Toll-Free Analysis

Safety Endpoints: Percentage of subjects occurred solicited events from the start of administration of study medications before colonoscopy. Percentage of subjects with treatment-emergent adverse events during the study period.

Eligible participants will be randomly assigned in a 1:1 ratio to one of two groups: Advanced Bowel Preparation (Group A): Participants will receive a PLD along with an APP based educational platform ( Tian Tian Yi Chi go) and Traditional Bowel Preparation (Group B).

Subject Population Assuming an acceptable bowel preparation rate of 70% for Traditional Bowel Preparation and 90% for Advanced Bowel Preparation, a significance level (α) of 0.05, statistical power of 80%, Single tailed test, and accounting for a 10% dropout rate, approximately 207 subjects per group (total 420 subjects) are required.

Inclusion Criteria Male or female 18 to 75 years of age. Bowklean naive patient with no bowel preparation in 3 years. The subject is scheduled for a colonoscopy. Ability to complete the entire procedure and to comply with study instructions. Willingness and ability to provide signed informed consent.

Exclusion Criteria Patients who are unsuitable for Bowklean use due to known contraindications, including but not limited to: (1) Allergies or hypersensitivity to Bowklean or its ingredients. (2) Severe gastrointestinal conditions (e.g., obstruction, perforation). (3) Renal impairment or electrolyte imbalances (e.g., severe hyponatremia). (4) Gastrointestinal surgery affects bowel preparation. Patients deemed medically unsuitable for colonoscopy by the physician. Cognitive, language, or other barriers that prevent completion of the questionnaire. Non-compliance with the bowel preparation protocol or inability to follow dietary restrictions (e.g., Prepackaged low residue diet, PLD). Inability to use or access the mobile APP (e.g., no smartphone, unfamiliarity with APP operations, or technical limitations). Participation in other clinical trials.

Discontinuation Criteria of Subjects Discontinuation is a subject who is randomized into the study and for whom study medication (Group A or Group B) is terminated prematurely for any reason. The subject is free to withdraw from the study for any reason and at any time without giving reason for doing so and without penalty or prejudice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 75 years of age.
2. Bowklean naive patient with no bowel preparation in 3 years.
3. The subject is scheduled for a colonoscopy.
4. Ability to complete the entire procedure and to comply with study instructions.
5. Willingness and ability to provide signed informed consent.

Exclusion Criteria:

1. Patients who are unsuitable for Bowklean use due to known contraindications, including but not limited to:

1. Allergies or hypersensitivity to Bowklean or its ingredients.
2. Severe gastrointestinal conditions (e.g., obstruction, perforation).
3. Renal impairment or electrolyte imbalances (e.g., severe hyponatremia).
4. Gastrointestinal surgery affects bowel preparation. 2. Patients deemed medically unsuitable for colonoscopy by the physician. 3. Cognitive, language, or other barriers that prevent completion of the questionnaire.

4. Non-compliance with the bowel preparation protocol or inability to follow dietary restrictions (e.g., Prepackaged low residue diet, PLD).

5. Inability to use or access the mobile APP (e.g., no smartphone, unfamiliarity with APP operations, or technical limitations).

6. Participation in other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-10-21 (Estimated); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects that achieve adequate cleansing | Day1
  The percentage of subjects that achieve adequate cleansing (score ≧ 6) in the Boston Bowel Preparation Scale (BBPS)

SECONDARY OUTCOMES:
The percentage of subjects that achieve excellent cleansing | Day1
  (score ≧ 8) in the Boston Bowel Preparation Scale (BBPS).
Mean score in different colon segments | Day1
  right, transverse, left colon segmental subscore, which are assessed with the BBPS.
Adenoma Detection Rate (ADR) | Day14
  Proportion of patients in whom at least one adenoma is detected during the colonoscopy.
Sessile Serrated Polyp (SSP) Detection Rate | Day14
  Proportion of patients in whom at least one SSP is detected during the colonoscopy.
Patient Satisfaction | Day1
  Satisfaction will be evaluated in three subcategories through a questionnaire:
  1. Bowel cleansing agent: Assessing the experience and acceptability of using Bowklean.
  2. Dietary restrictions: Evaluating satisfaction with the assigned low-residue dietary approach (PLD or self-prepared).
  3. APP Satisfaction: For groups assigned to APP utilization, assessing the APP's ease of use, functionality, and perceived utility.